CLINICAL TRIAL: NCT00075413
Title: A Pilot Phase II Protocol Of Arsenic Trioxide (TRISENOX) In Subjects With Advanced Carcinoma Of The Breast
Brief Title: Arsenic Trioxide in Treating Women With Locally Advanced or Metastatic Breast Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Unable to identify qualified subjects willing to participate in this study
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000346365; UTMB-02403
Record Dates: First submitted 2004-01-09; First posted 2004-01-12 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-09

CONDITIONS: Breast Cancer
Keywords: stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Arsenic Trioxide

INTERVENTIONS:
Drug: arsenic trioxide

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as arsenic trioxide, use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: This phase II trial is studying how well arsenic trioxide works in treating women with locally advanced or metastatic breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the safety and activity of arsenic trioxide in women with locally advanced or metastatic breast cancer.
* Determine the qualitative and quantitative toxic effects of this drug in these patients.

Secondary

* Determine the response, in terms of objective tumor response and response duration, in patients treated with this drug.
* Determine the patterns of failure and survival in patients treated with this drug.

OUTLINE: This is a pilot study.

Patients receive arsenic trioxide IV over 1-2 hours on days 1-5 of week 1 and on days 1 and 5 of weeks 2-8 (for course 1 only). Beginning with course 2 and for all subsequent courses, patients receive arsenic trioxide on days 1 and 5 of weeks 1-8. Treatment repeats every 8 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Patients who have a complete response (CR) receive an additional course beyond documentation of CR. Patients who have a CR due to local consolidative therapy (e.g., surgery or radiotherapy) receive an additional 2 courses beyond CR.

Patients are followed for 1 month, every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 14-30 patients will be accrued for this study within 9-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed breast cancer, meeting 1 of the following criteria:

  * Locally advanced disease

    * Cannot be adequately treated by radiotherapy or surgery
  * Metastatic disease
* Ineligible for OR received prior anthracycline- and/or taxane-based chemotherapy with subsequent disease progression
* No uncontrolled Central Nervous System (CNS) metastases
* Ineligible for treatment protocols of higher priority
* Hormone receptor status:

  * Not specified

PATIENT CHARACTERISTICS:

Age

* 18 and over

Sex

* Female

Menopausal status

* Not specified

Performance status

* Eastern Cooperative Oncology Group (ECOG) 0-1 OR
* Southwest Oncology Group (SWOG) 0-1 OR
* Zubrod 0-1

Life expectancy

* At least 12 weeks

Hematopoietic

* Absolute neutrophil count greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic

* Bilirubin no greater than 1.5 times normal
* Serum Glutamic Oxalacetic Transaminase (SGOT)/Serum Glutamic Pyruvic Transaminase (SGPT) no greater than 3 times normal

Renal

* Creatinine no greater than 2.0 mg/dL
* Calcium no greater than 12 mg/dL

Cardiovascular

* Cardiac ejection fraction greater than 50%
* No myocardial infarction or ischemia within the past 6 months
* No uncontrolled clinically significant dysrhythmia

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* Electrolytes normal
* Magnesium normal
* No other malignancy within the past 5 years except nonmelanoma skin cancer or carcinoma in situ of the cervix
* No prior or ongoing grade 2-4 peripheral neuropathy
* No comorbid condition that would render the patient at high risk from study treatment complications

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No concurrent cytokine therapy

Chemotherapy

* See Disease Characteristics
* No more than 3 prior chemotherapy regimens for breast cancer
* No other concurrent chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* More than 2 weeks since prior radiotherapy
* No prior radiotherapy to an indicator lesion unless there is objective evidence of tumor growth in that lesion
* No concurrent radiotherapy except for the following:

  * Palliative or emergent radiotherapy
  * Local consolidative radiotherapy

Surgery

* More than 2 weeks since prior surgery
* Concurrent local consolidative surgery allowed

Other

* At least 4 weeks since prior antineoplastic agents for nonmalignant conditions (e.g., methotrexate for rheumatoid arthritis)
* No concurrent antineoplastic agents for nonmalignant conditions
* No concurrent participation in another treatment protocol
* Concurrent local palliative therapy allowed

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2002-11; Primary Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennie V. Jones, MD, Study Chair — University of Texas